CLINICAL TRIAL: NCT00758602
Title: A Randomized, Open Label Study Comparing the Effect of CellCept Combined With Low Dose Versus Standard Dose Tacrolimus, and Corticosteroids, on Kidney Function in Renal Transplantation Patients
Brief Title: A Study of CellCept (Mycophenolate Mofetil) Combined With Tacrolimus and Corticosteroids in Kidney Transplant Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21740
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Tacrolimus; Adrenal Cortex Hormones

ARMS (2):
- MMF, Standard Dose Tacrolimus (Active Comparator): Participants received mycophenolate mofetil (MMF) 0.75 to (-) 1 gram (g), orally (PO), twice daily (BID) from Day 0 through Month 12. Participants also received tacrolimus 0.1-0.15 milligrams per kilogram (mg/kg), PO, BID to reach a target trough dose of 8-10 nanograms per milliliter (ng/mL) from Day 0 through Month 3; the dose was adjusted to reach a target trough level of 7-10 ng/mL in Month 3 and continued through Month 12. Participants also received corticosteroids per center practice.
  Interventions: Drug: mycophenolate mofetil; Drug: tacrolimus, standard dose; Drug: corticosteroids
- MMF, Low Dose Tacrolimus (Experimental): Participants received MMF 0.75-1 g, PO, BID from Day 0 through Month 12. Participants also received tacrolimus 0.1-0.15 mg/kg, PO, BID to reach a target trough dose of 8-10 ng/mL from Day 0 through Month 3; the dose was adjusted to 0.05-0.08 mg/kg, PO, BID to reach a target trough dose of 2-5 ng/mL in Month 3 and continued through Month 12. Participants also received corticosteroids per center practice.
  Interventions: Drug: mycophenolate mofetil; Drug: tacrolimus, low dose; Drug: corticosteroids

INTERVENTIONS:
Drug: mycophenolate mofetil — 0.75-1 g PO BID from Day 0 through Month 12
  Other Names: CellCept
Drug: tacrolimus, standard dose — Initial dose of 0.1-0.15 mg/kg PO BID to reach a target trough dose of 8-10 ng/mL from Day 0 through Month 3; the dose was adjusted to reach a target trough level of 7-10 ng/mL in Month 3 and continued through Month 12.
  Arms: MMF, Standard Dose Tacrolimus
Drug: tacrolimus, low dose — Initial dose of 0.1-0.15 mg/kg PO BID to reach a target trough dose of 8 to 10 ng/mL from Day 0 through Month 3; 0.05-0.08 mg/kg PO BID to reach a target trough dose of 2-5 ng/mL in Month 3 and continued through Month 12.
  Arms: MMF, Low Dose Tacrolimus
Drug: corticosteroids — According to center's practice

SUMMARY:
This 2 arm study will compare the efficacy and safety of CellCept, combined with low or standard dose tacrolimus plus corticosteroids, in patients with kidney transplants. Patients will be randomized into one of 2 groups to receive either 1)CellCept 2.0g/day po bid + tacrolimus 10-12ng/mL followed by a maintenance dose of 8-10ng/mL + corticosteroids or 2)CellCept 2.0g/day po bid + tacrolimus 8-10ng/mL in the first 2 months,3-7ng/mL in month 3 followed by a maintenance dose of 3-5ng/mL + corticosteroids. The anticipated time on study treatment is 1 year, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, <=75 years of age;
* single organ recipients of renal allograft;
* negative pregnancy test for women of childbearing potential; reliable contraception must be used before starting drug therapy, until 6 weeks after the last dose of study medication.

Exclusion Criteria:

* severe gastrointestinal disease which may influence the absorption of oral drug therapy;
* severe infection, HIV or active hepatitis;
* active gastric ulcers;
* malignancy other than cured skin cancer;
* severe anemia, leucopenia or thrombocytopenia.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- China (6):
  - Beijing
  - Fuzhou
  - Guangzhou
  - Nanjing
  - Shanghai
  - Zhejiang

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil (MMF), Standard Dose Tacrolimus: Participants received MMF capsules, 0.75-1 gram (g) orally (PO), twice daily (BID) from Day 0 through Month 12 (maximum dose administered was 1.5 g BID, at discretion of investigator). Participants also received tacrolimus PO, BID, dosed to reach a target trough level of 10-12 nanograms per milliliter (ng/mL) from Day 0 through Month 3; the dose was adjusted to reach a target trough level of 8-10 ng/mL in Month 3 and continued through Month 12. Participants also received intraoperative and maintenance corticosteroids per center practice.
- MMF, Low Dose Tacrolimus: Participants received MMF capsules, 0.75-1 g PO, BID from Day 0 through Month 12 (maximum dose administered was 1.5 g BID, at discretion of investigator. Participants also received tacrolimus PO, BID, dosed to reach a target trough level of 8-10 ng/mL from Day 0 through Month 2; the dose was adjusted reach a target trough level of 3-7 ng/mL in Month 3 and adjusted to achieve a target trough level of 3-5 ng/mL thereafter, through Month 12. Participants also received intraoperative and maintenance corticosteroids per center practice.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF), Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Started | 104 | 106
Completed | 85 | 84
Not Completed | 19 | 22
Not completed — Adverse Event | 11 | 10
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 0 | 1
Not completed — Reason not specified | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all randomized patients who received at least one dose ofthe treatment-group specific medication.
Groups:
- MMF, Standard Dose Tacrolimus: Participants received MMF capsules, 0.75-1 g PO, BID from Day 0 through Month 12 (maximum dose administered was 1.5 g BID, at discretion of investigator). Participants also received tacrolimus PO, BID, dosed to reach a target trough level of 10-12 ng/mL from Day 0 through Month 3; the dose was adjusted to reach a target trough level of 8-10 ng/mL in Month 3 and continued through Month 12. Participants also received intraoperative and maintenance corticosteroids per center practice.
- Total: Total of all reporting groups
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus | Total
Number analyzed (Participants) | 104 | 106 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (11.05) | 39.6 (10.16) | 38.8 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 75 | 72 | 147

OUTCOME MEASURES:

1. Primary Outcome: Chronic Allograft Damage Index (CADI) Score at Month 12 After Transplantation
Description: CADI scoring was defined for 6 histological categories: interstitial inflammatory cell infiltration (0 equals (=) no or mild inflammation, 1=approximately (~)25 percent (%) cell infiltration, 2=26-50% cell infiltration, and 3=greater than (>)50% cell infiltration); interstitial fibrosis (0=none, 1=~25% interstitial affected, 2=26-50% interstitial affected, and 3=>50% interstitial affected); tubular atrophy (0=none, 1=~15% proximal tubular atrophy [PTA], 2=16-30% PTA, and 3=>30% PTA); mesangial matrix proliferation (MMP; 0=none, 1=25% non-glomerulosclerosis [NGS] combined with moderate MMP, 2=25-50% NGS combined with MMP, and 3=>50% NGS combined with MMP); glomerular sclerosis (0=none, 1=~15% glomerulus affected, 2=16-50% glomerulus affected, and 3=>50% glomerulus affected); endothelial proliferation (EP; 0=none, 1=EP to less than (<)25% remaining artery/small artery membrane [RA/SAM], 2=EP to 26-50% [RA/SAM], and 3=>50% [RA/SAM]). CADI score was the sum of the 6 histological findings.
Time Frame: Month 12
Population: ITT population; only participants with biopsy confirmed CADI assessment 12 months post-transplantation were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 57 | 52
score on a scale | 1.82 (1.974) | 2.13 (2.000)
Statistical Analysis 1: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Test type: Superiority or Other; p = 0.0813, ANCOVA — p-value, least squares (LS) mean difference, and 95% confidence interval (CI) based on analysis of covariance (ANCOVA) model with treatment, center, and the treatment-by-center interaction as fixed effects, and the donor age as a covariate; LS Mean difference = 0.6581, 95% CI 2-sided [-0.08 to 1.40]

2. Primary Outcome: Glomerular Filtration Rate (GFR) at Month 12 After Transplantation
Description: GFR was determined using the Cockcroft-Gault formula to calculate the creatinine clearance, at Month 12 after renal transplantation. For males, creatinine clearance [milliliters per minute (mL/min)] = [(140 minus age) multiplied by (*) (body weight in kg) divided by [72 * serum creatinine mg per deciliter (mg/dL)]. For females, creatinine clearance (mL/min) = 0.85 * [(140 minus age) * (body weight in kg)] divided by [72 * serum creatinine (mg/dL)].
Time Frame: Month 12
Population: ITT population; only participants with assessable parameters for the calculation of GFR were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 86 | 82
mL/min | 77.08 (18.250) | 80.12 (18.362)
Statistical Analysis 1: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Test type: Superiority or Other; p = 0.7949, ANCOVA — p-value, LS mean difference, and 95% CI based on ANCOVA model with treatment, center, and the treatment-by-center interaction as fixed effects, and the donor age as a covariate; LS Mean difference = -1.5977, 95% CI 2-sided [-13.77 to 10.58]

3. Secondary Outcome: Percentage of Participants Experiencing Acute Rejection, Graft Loss, or Death at 6 and 12 Months Post-Transplant
Time Frame: Months 6 and 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
percentage of participants
  Acute rejection, 6 months post-transplant | 2.6 | 5.2
  Acute rejection, 12 months post-transplant | 2.6 | 5.2
  Graft loss, 6 months post-transplant | 0.0 | 0.0
  Graft loss, 12 months post-transplant | 0.0 | 0.0
  Death, 6 months post-transplant | 0.0 | 0.0
  Death, 12 months post-transplant | 0.0 | 0.9
Statistical Analysis 1: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Acute rejection, 6 months post-transplant; Test type: Superiority or Other; p = 0.6812, Fisher Exact
Statistical Analysis 2: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Acute rejection, 12 months post-transplant; Test type: Superiority or Other; p = 0.6812, Fisher Exact
Statistical Analysis 3: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Death, 12 months post-transplant; Test type: Superiority or Other; p = 1.0000, Fisher Exact

4. Secondary Outcome: Time to First Acute Rejection Post-Transplant - Number of Participants With an Event
Time Frame: BL, Weeks 2, 4, 13, 26, 39, and 52
Population: ITT population
Measure: Number; unit: participants
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
participants | 2 | 4

5. Secondary Outcome: Time to First Acute Rejection Post-Transplant
Description: The median time, in days, between randomization and acute rejection.
Time Frame: BL, Weeks 2, 4, 13, 26, 39, and 52
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
days | 40 [13 to 67] | 18 [5 to 95]
Statistical Analysis 1: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Test type: Superiority or Other; p = 1.0000, Log Rank

6. Secondary Outcome: Percentage of Participants With Treatment Failure at 12 Months Post-Transplant
Description: Treatment failure was defined by the occurrence of any of the following: use of additional maintenance immunosuppressive medication not specified in the assigned treatment group; discontinuation of any of the assigned immunosuppressants for more than 14 consecutive days or 30 cumulative days; graft loss or return to chronic dialysis; or death.
Time Frame: Month 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
percentage of participants | 9.6 | 6.6
Statistical Analysis 1: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Test type: Superiority or Other; p = 0.4586, Fisher Exact

7. Secondary Outcome: Participant and Graft Survival
Description: The percentage of participants surviving with grafts intact at 6 and 12 months after renal transplant.
Time Frame: Months 6 and 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
percentage of participants
  6 months post-transplant | 100.0 | 100.0
  12 months post-transplant | 100.0 | 99.1
Statistical Analysis 1: Comparison: MMF, Standard Dose Tacrolimus vs MMF, Low Dose Tacrolimus; Test type: Superiority or Other; p = 1.0000, Fisher Exact

8. Secondary Outcome: Serum Creatinine (Micromoles Per Liter [µmol/L])
Description: The mean serum creatinine values in µmol/L at Baseline (BL), Weeks 2, 4, 13, 26, 39, and 52.
Time Frame: BL, Weeks 2, 4, 13, 26, 39, and 52
Population: ITT population; n (number) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- MMFl, Low Dose Tacrolimus: Participants received MMF capsules, 0.75-1 g PO, BID from Day 0 through Month 12 (maximum dose administered was 1.5 g BID, at discretion of investigator. Participants also received tacrolimus PO, BID, dosed to reach a target trough level of 8-10 ng/mL from Day 0 through Month 2; the dose was adjusted reach a target trough level of 3-7 ng/mL in Month 3 and adjusted to achieve a target trough level of 3-5 ng/mL thereafter, through Month 12. Participants also received intraoperative and maintenance corticosteroids per center practice.
Arm/Group | MMF, Standard Dose Tacrolimus | MMFl, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
µmol/L
  Baseline (n=95,96) | 662.93 (351.913) | 639.70 (287.044)
  Week 2 (n=101,102) | 154.57 (151.374) | 115.71 (52.648)
  Week 4 (n=99,98) | 118.47 (76.134) | 107.08 (32.668)
  Week 13 (n=88,91) | 97.52 (24.947) | 100.10 (25.345)
  Week 26 (n=84,83) | 105.70 (45.403) | 97.51 (21.997)
  Week 39 (n=83,77) | 102.22 (38.035) | 95.16 (20.877)
  Week 52 (n=86,82) | 103.10 (48.251) | 94.19 (21.964)

9. Secondary Outcome: Glomerular Filtration Rate (GFR) (mL/Min)
Description: The mean GFR values in mL/min at BL, Weeks 2, 4, 13, 26, 39, and 52.
Time Frame: BL, Weeks 2, 4, 13, 26, 39, and 52
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Number analyzed (Participants) | 104 | 106
mL/min
  Baseline (n=95,96) | 14.37 (8.080) | 15.41 (13.759)
  Week 2 (n=101,102) | 67.95 (30.140) | 71.02 (22.177)
  Week 4 (n=99,98) | 71.77 (23.578) | 72.87 (19.934)
  Week 13 (n=88,91) | 78.13 (18.686) | 75.71 (17.906)
  Week 26 (n=84,83) | 75.92 (21.046) | 76.77 (17.536)
  Week 39 (n=83,77) | 77.34 (19.046) | 78.00 (16.036)
  Week 52 (n=86,82) | 77.08 (18.250) | 80.12 (18.362)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from study start to 1 month after treatment completion. Treatment related serious AEs (SAEs) were reported no matter how long after the last treatment dose was administered, even though the study had been terminated.
Description: All randomized participants were included in the safety analysis.
Arm/Group | MMF, Standard Dose Tacrolimus | MMF, Low Dose Tacrolimus
Serious Adverse Events (participants affected / at risk) | 1/104 | 5/106
Other Adverse Events (participants affected / at risk) | 33/104 | 37/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF, Standard Dose Tacrolimus (N=104) | MMF, Low Dose Tacrolimus (N=106)
Sudden death (Cardiac disorders) | 0 | 1
Acute rejection (Renal and urinary disorders) | 1 | 1
Transplanted renal rupture (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Cytomegalovirus (CMV) disease (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF, Standard Dose Tacrolimus (N=104) | MMF, Low Dose Tacrolimus (N=106)
Alanine transaminase (ALT) increased (Investigations) | 10 | 12
White blood cell (WBC) count decreased (Blood and lymphatic system disorders) | 9 | 9
Diarrhea (Gastrointestinal disorders) | 4 | 8
Serum creatinine increased (Renal and urinary disorders) | 5 | 4
Aspartate transamininase (AST) increased (Investigations) | 4 | 3
Hyperlipemia (Investigations) | 3 | 4
New-onset diabetes (Endocrine disorders) | 3 | 2
Pyrosis (Gastrointestinal disorders) | 0 | 4
Nausea/vomiting (Gastrointestinal disorders) | 1 | 1
Hypercholesterolemia (Investigations) | 1 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1 | 0
Others - not specified (General disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.